CLINICAL TRIAL: NCT05890885
Title: The Effect of Home-Based Transcranial Direct Current Stimulation on Fatigue in Multiple Sclerosis
Brief Title: MS Fatigue and tDCS on Fatigue in Multiple Sclerosis
Acronym: MSfatDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: APHP210747
Record Dates: First submitted 2022-01-05; First posted 2023-06-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fatigue in Multiple Sclerosis
Keywords: Fatigue; Multiple sclerosis; Anodal tDCS; Prefrontal cortex
MeSH Terms: conditions — Fatigue; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: During a routine visit in the Department of Neurology for monitoring MS disease, patients undergo a routine neurological exam which will serve later on to check inclusion/exclusion criteria (i.e., this exam will help rating the disability using the Expanded Disability Status Scale that is also routinely performed in all patients with MS). If a patient is interested in this research, the information form will be given to him/her by one of the study investigators (screening visit).
  Then, after a period of reflection of at least one week after the screening visit, one study investigator will call the patient to inquire about her/his willingness to participate to the study. If the patient agrees to participate in this research, (s)he will be invited for a baseline visit in the Department of Clinical Neurophysiology for inclusion in the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real - Sham (Experimental): Real left prefrontal tDCS followed by sham tDCS after a 4-week washout period
  Interventions: Procedure: Real left prefrontal tDCS - sham
- Sham - Real (Experimental): Sham tDCS followed by real left prefrontal tDCS after a 4-week washout period
  Interventions: Procedure: Sham - Real left prefrontal tDCS

INTERVENTIONS:
Procedure: Real left prefrontal tDCS - sham — Real left prefrontal tDCS followed by sham tDCS after a 4-week washout period
  Arms: Real - Sham
Procedure: Sham - Real left prefrontal tDCS — Sham tDCS followed by real left prefrontal tDCS after a 4-week washout period
  Arms: Sham - Real

SUMMARY:
The available therapeutic strategies for Multiple Sclerosis (MS)-related symptoms are usually faced with limited efficacy and numerous side effects. Patients with MS frequently suffer from fatigue, affective symptoms, and cognitive deficits.

DETAILED DESCRIPTION:
For these reasons, non-invasive brain stimulation (NIBS) techniques, namely transcranial direct current stimulation (tDCS) might be of help in this context. tDCS is a new NIBS technique with a good safety profile, easy implementation, good patients' tolerance and little or no adverse effects. tDCS uses low levels of constant current delivered to specific brain area via sponge electrodes placed on the scalp. tDCS modifies the polarization of the exposed neuronal circuits. Indeed, it modulates the spontaneous neuronal excitability and activity by a tonic depolarization or hyperpolarization of resting membrane potential.

Therefore, applying a home-based intervention is of interest in a population suffering from high levels of physical disability prohibiting them from frequently coming to seek care at the hospital

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis according to the 2017 McDonald criteria
* Fatigue since more than 6 months as assessed by fatigue severity scale (FSS>5)
* Age between 18 and 75 years.
* Stable pharmacological and physical treatment since at least one month
* Affiliation to the social security regimen
* Signature of the informed consent
* Ability of the patient to understand the instructions for use of the pacemaker to ensure safe use

Exclusion Criteria:

* Relapses within the last two months
* Active medical device implanted
* Intracranial metal implants
* Craniotomy, cranial trepanation, aneurysm
* Uncontrolled epilepsy
* Non-weaned alcoholism, sleep debt
* Expanded disability status scale ≥ 6.5
* Severe depression based on Beck Depression inventory (BDI>19)
* Daytime sleepiness based on Epworth Sleepiness Scale (ESS> 11)
* Other neurologic and psychiatric diseases
* Known pregnancy by the investigator or breastfeeding
* Physical or mental incapacity to give informed consent
* Participation in another study (exclusion period following a previous study should be ≥ 6 months)
* Patients on AME
* Patients under legal protection
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Tiredness | 12 weeks
  Modified Fatigue Impact Scale (MFIS): cognitive (10 items), physical (9 items) and psychosocial fatigue (2 items). It is a shortened version of the Fatigue Impact Scale that contains 21 of the original 40 items.

SECONDARY OUTCOMES:
Depression | 12 weeks
  Mood will be assessed by the Hospital Anxiety and Depression Scale (HADS), which is composed of 7 questions that assess anxiety and 7 questions that assess depression.
Anxiety | 12 weeks
  Mood will be assessed by the Hospital Anxiety and Depression Scale (HADS), which is composed of 7 questions that assess anxiety and 7 questions that assess depression.
Alexithymia | before and after each stimulation period (active and simulated) and four weeks later (four weeks after the last stimulation session of each period).
  Alexithymia will be assessed using the 20-item Toronto Alexithymia Scale (TAS), which assesses the difficulties in analysing and describing one's own feelings and an externally oriented thinking.
MSQOL scale | 12 weeks
  Quality of life will be assessed using the MS quality of life questionnaire (MSQOL), which is a multidimensional scale that assess different functions and can yield physical and mental composite scores.
Cognitive functions | 12 weeks
  Cognitive functions will be assessed using the cognitive domain of the MSQOL, the Reading the Mind in the Eyes Test (RMET) and empathy quotient (EQ), which evaluated social cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Samar AYACHE, Principal Investigator — Clinical Neurophysiology Department
Locations (1):
- Assistance Publique Hôpitaux de Paris-Hôpital Henri Mondor, Créteil, France